CLINICAL TRIAL: NCT03927430
Title: To Peel or Not to Peel: Surgical Outcome of Macular Membrane Peeling Associated With Significant Macular Drusen
Brief Title: Surgical Outcome of Macular Membrane Peeling Associated With Significant Macular Drusen
Status: Completed | Type: Observational
Sponsor: Klinikum Chemnitz gGmbH (Other)
Responsible Party: Principal Investigator, Katrin Engelmann, Head of Ophthalmology, Klinikum Chemnitz gGmbH
Other Study IDs: SKC01/2019
Record Dates: First submitted 2019-04-15; First posted 2019-04-25 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Epiretinal Membrane; Macular Holes; Age Related Macular Degeneration
MeSH Terms: conditions — Epiretinal Membrane; Retinal Perforations; Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pars plana vitrectomy with membrane peeling — 23-gauge pars plana vitrectomy with peeling of the epiretinal and internal limiting membrane as well as air- or gastamponade

SUMMARY:
Surgical outcome of patients with macular drusen and co-existing abnormalities of the vitreoretinal interface, who routinely undergo pars plana vitrectomy with membrane peeling, is evaluated. Best corrected visual acuity as well as optical coherence tomography data are compared at baseline and last follow up. The rate of development of choroidal neovascularization postoperatively is noted.

ELIGIBILITY:
Inclusion Criteria:

1. participants diagnosed with ERM or FTMH and co-existing macular drusen;
2. undergone pars plana vitrectomy with ILM and epiretinale membrane peeling;
3. SD-OCT at the initial visit and at last follow up visit with image quality score >30;
4. no evidence of CNV on initial fluorescein angiography (FA).

Exclusion Criteria:

1. history of other macular disease, severe non-proliferative or proliferative diabetic retinopathy, other retinal vascular diseases, glaucoma, myopic retinopathy, or other diseases interfering with OCT images in any one of the eyes;
2. active CNV or history of CNV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mostly elderly people, mean age 66 years, both males and females
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
number of patients with CNV | last visit, in common 6 months postoperatively
  number of patients with CNV (choroidal neovascularization) development

SECONDARY OUTCOMES:
BCVA | last visit, in common 6 months postoperatively
  best corrected visual acuity
incidence of central retinal atrophy | last visit, in common 6 months postoperatively
  development of central retinal atrophy on OCT

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Engelmann, PhD, Study Chair — Klinikum Chemnitz
Locations (1):
- Klinikum Chemnitz, Ophthalmology Department, Chemnitz, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No